CLINICAL TRIAL: NCT00073658
Title: Continuation Pharmacotherapy for Agitation of Dementia
Brief Title: Treating Behavioral Disturbances in Individuals With Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH059666-02 (NIH); R01MH059666-02 (NIH); DSIR GT-GP
Record Dates: First submitted 2003-12-02; First posted 2003-12-03 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Dementia
Keywords: Alzheimer disease; Aggression; Delusions; Paranoid behavior
MeSH Terms: conditions — Dementia; Alzheimer Disease; Aggression; Delusions; Paranoid Behavior | interventions — Citalopram; Risperidone

INTERVENTIONS:
Drug: Citalopram
Drug: Risperidone

SUMMARY:
This study will compare the safety and effectiveness two medications, citalopram (Celexa®) and risperidone (Risperdal®).

DETAILED DESCRIPTION:
Dementia-related behavioral disturbances have been associated with excess disability, increased caregiver burden, and premature institutionalization. Pharmacotherapy is often necessary to treat these disturbances. This study will use citalopram and risperidone to treat people with dementia-related behavior problems.

Participants in this study will begin a psychotropic medication washout period for up to 3 days at study start. Participants will then be randomly assigned to receive either citalopram or risperidone for up to 12 weeks. Limited doses of the sedative lorazepam may be administered as needed throughout the study. During the first 2 weeks of the study, participants will be admitted to a hospital to have their dementia-related behavioral disturbances stabilized. Following hospital discharge, participants will move to a long-term care facility or a residential home and will continue medication treatment for up to 10 weeks. Side effects and improvements in behavioral status will be assessed every week until Week 6 and every 2 weeks thereafter. Experimental laboratory measures will be collected at study start, Week 1, Week 2, and every 2 weeks thereafter until Week 12. Upon study completion, patients may continue to receive citalopram or risperidone under the supervision of their current physicians. Three months after study completion, participants may be contacted for a follow-up report of their psychiatric and medical status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's type dementia and/or meet criteria for probable or possible Alzheimer's disease
* Inpatient admittance to Western Psychiatric Institute and Clinic
* Written informed consent from participant's legally authorized representative with the participant's assent
* Psychosis or behavioral problems severe enough to be a danger to the participant's health, well-being, or safety
* Score of 3 to 6 (moderate to severe) on at least one of the Neurobehavioral Rating Scale (NBRS) agitation or psychosis items
* Ability to participate in study evaluation and ingest oral medication

Exclusion Criteria:

* Diagnosis of an unstable medical illness within the last 12 months
* Kidney or liver dysfunction
* Diagnosis of delirium, substance-induced persisting dementia, or vascular dementia
* Score of 12 or higher on the Cornell Scale for Depression in Dementia, and a score greater than 3 on the depression item of the NBRS
* Diagnosis of Parkinson's disease or any neurological illness which may affect cognitive function
* History of schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, or bipolar affective disorder
* Alcohol or substance abuse or dependence
* Receiving monoamine oxidase inhibitors within 15 days of study
* Display behaviors which could endanger the participant's life or the lives of others
* Received fluoxetine within 4 weeks of screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137
Dates: Start 2000-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Pollock, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center/Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Sweet RA, Pollock BG, Sukonick DL, Mulsant BH, Rosen J, Klunk WE, Kastango KB, DeKosky ST, Ferrell RE. The 5-HTTPR polymorphism confers liability to a combined phenotype of psychotic and aggressive behavior in Alzheimer disease. Int Psychogeriatr. 2001 Dec;13(4):401-9. doi: 10.1017/s1041610201007827. PMID 12003247
- [Background] Maxwell RA, Sweet RA, Mulsant BH, Rosen J, Kirshner MA, Kastango KB, Pollock BG. Risperidone and 9-hydroxyrisperidone concentrations are not dependent on age or creatinine clearance among elderly subjects. J Geriatr Psychiatry Neurol. 2002 Summer;15(2):77-81. doi: 10.1177/089198870201500205. PMID 12083597
- [Background] Carnahan RM, Lund BC, Perry PJ, Pollock BG. A critical appraisal of the utility of the serum anticholinergic activity assay in research and clinical practice. Psychopharmacol Bull. 2002 Spring;36(2):24-39. PMID 12397838
- [Background] Mamo DC, Sweet RA, Mulsant BH, Rosen J, Pollock BG: Neuroleptic-induced Parkinsonism in Alzheimer's disease. Psychiatric Annals 32:249-252, 2002.
- [Background] Pollock BG, Mulsant BH, Rosen J, Sweet RA, Mazumdar S, Bharucha A, Marin R, Jacob NJ, Huber KA, Kastango KB, Chew ML. Comparison of citalopram, perphenazine, and placebo for the acute treatment of psychosis and behavioral disturbances in hospitalized, demented patients. Am J Psychiatry. 2002 Mar;159(3):460-5. doi: 10.1176/appi.ajp.159.3.460. PMID 11870012
- [Background] Kastango KB, Kim Y, Dew MA, Mazumdar S, Mulsant BH, Rosen J, Reynolds III CF, Pilkonis PA, Pollock BG. Verification of scale sub-domains in elderly patients with dementia: a confirmatory factor-analytic approach. Am J Geriatr Psychiatry. 2002 Nov-Dec;10(6):706-14. PMID 12427579
- [Background] Bies RR, Gastonguay MR, Coley KC, Kroboth PD, Pollock BG. Evaluating the consistency of pharmacotherapy exposure by use of state-of-the-art techniques. Am J Geriatr Psychiatry. 2002 Nov-Dec;10(6):696-705. PMID 12427578
- [Background] Mulsant BH, Pollock BG, Kirshner M, Shen C, Dodge H, Ganguli M. Serum anticholinergic activity in a community-based sample of older adults: relationship with cognitive performance. Arch Gen Psychiatry. 2003 Feb;60(2):198-203. doi: 10.1001/archpsyc.60.2.198. PMID 12578438
- [Background] Bharucha AJ, Rosen J, Mulsant BH, Pollock BG. Assessment of behavioral and psychological symptoms of dementia. CNS Spectr. 2002 Nov;7(11):797-802. doi: 10.1017/s1092852900024317. PMID 12947242
- [Background] Lotrich FE, Pollock BG, Ferrell RE. Serotonin transporter promoter polymorphism in African Americans : allele frequencies and implications for treatment. Am J Pharmacogenomics. 2003;3(2):145-7. doi: 10.2165/00129785-200303020-00007. PMID 12749731
- [Derived] Culo S, Mulsant BH, Rosen J, Mazumdar S, Blakesley RE, Houck PR, Pollock BG. Treating neuropsychiatric symptoms in dementia with Lewy bodies: a randomized controlled-trial. Alzheimer Dis Assoc Disord. 2010 Oct-Dec;24(4):360-4. doi: 10.1097/WAD.0b013e3181e6a4d7. PMID 20625270